CLINICAL TRIAL: NCT03966118
Title: Avelumab + Paclitaxel/ Ramucirumab as Second Line Treatment in Gastro-esophageal Adenocarcinoma: a Phase II Trial of the AIO (The RAP-Trial)
Brief Title: Avelumab + Paclitaxel/ Ramucirumab (RAP) as Second Line Treatment in Gastro-esophageal Adenocarcinoma
Acronym: AIO-STO-0218
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: P. C. Thuss-Patience (Other)
Responsible Party: Sponsor-Investigator, P. C. Thuss-Patience, MD (Principal Investigator), Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAP-Trial
Record Dates: First submitted 2019-02-12; First posted 2019-05-29 (Actual); Last update posted 2019-06-03 (Actual); Status verified 2019-05

CONDITIONS: Gastroesophageal Junction Adenocarcinoma; Adenocarcinoma of the Stomach
Keywords: 2nd line; Ramucirumab; Avelumab; Paclitaxel; gastric cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — avelumab; Ramucirumab; Paclitaxel

STUDY DESIGN:
Intervention Model Description: Avelumab + Paclitaxel / Ramucirumab
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ramucirumab + Avelumab + Paclitaxel (Experimental): Single-Arm
  Interventions: Drug: Avelumab; Drug: Ramucirumab; Drug: Paclitaxel

INTERVENTIONS:
Drug: Avelumab — Avelumab 1mg/kg Day 1 and Day 15 of a 28-day cycle
Drug: Ramucirumab — Ramucirumab 8mg/kg on Day 1 and Day 15 of a 28-day cycle
Drug: Paclitaxel — Paclitaxel 80mg/m2 on Day 1, Day 8 and Day 15 of a 28-day cycle

SUMMARY:
Avelumab + Paclitaxel/ Ramucirumab as second line treatment in gastro-esophageal adenocarcinoma following first-line therapy with platinum and fluoropyrimidine doublet with or without anthracycline, docetaxel or trastuzumab

DETAILED DESCRIPTION:
Patients with adenocarcinoma of the gastro-esophageal junction or the stomach who have documented progression after being treated with a 1st line chemotherapy which contained at least a platinum and 5-FU (5-Flourouracil)can be included. All patients will receive a standard second line therapy with paclitaxel and ramucirumab plus the investigational drug avelumab, a checkpoint inhibitor. Clinical and radiographic assessment will be performed regularly. Patients will be treated until disease progression, untolerable toxicity or withdrawal of consent.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent
2. Male or female ≥ 18 years of Age
3. Histologically proven gastric adenocarcinoma including adenocarcinoma of the esophagogastric junction
4. Metastatic or locally advanced disease, not amenable to potentially curative resection
5. Documented objective radiological or clinical disease progression during or within 6 months of the last dose of first-line platinum and fluoropyrimidine doublet with or without anthracycline, docetaxel or trastuzumab. Neoadjuvant/adjuvant treatment is not counted unless progression occurs <6 months after completion of the treatment. In these cases neoadjuvant/adjuvant treatment is counted as first line.
6. Measurable or non-measurable but evaluable disease determined using guidelines RECIST 1.1
7. Eastern Cooperative Oncology Group (ECOG) performance status 0-1
8. Life expectancy > 12 weeks
9. Adequate hematological, hepatic and renal functions:

   1. Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
   2. Platelet count ≥ 100 x 109/L
   3. Hemoglobin ≥ 9 g/dl (may have been transfused)
   4. Total bilirubin ≤ 1.5 times the upper limit of normal (ULN) and AST and ALT ≤ 2.5 x ULN in absence of liver metastases, or ≤ 5 x ULN in presence of liver metastases; AP ≤ 5 x ULN
   5. Estimated creatinine clearance ≥ 30 mL/min according to the Cockcroft-Gault formula (or local institutional standard method)
   6. Urinary protein ≤ 1+ on dipstick or routine urinalysis (UA; if urinedipstick or routine analysis is ≥ 2+, a 24-hour urine collection for protein must demonstrate < 1000 mg of protein in 24 hours to allow participation in this protocol)
   7. Adequate coagulation function as defined by International Normalized Ratio (INR) ≤ 1,5 ULN, and a partial thromboplastin time (PTT) ≤ 5 seconds above the ULN (unless receiving anticoagulation therapy). Patients receiving warfarin/phenprocoumon must be switched to low molecular weight heparin and have achieved stable coagulation profile prior to first dose of protocol therapy.
10. Women of child-bearing potential must have a negative urine or serum pregnancy test
11. Highly effective contraception for both male and female subjects throughout the study and for at least 30 days after last avelumab and at least 3 months after last ramucirumab treatment administration if the risk of conception exists
12. Ability to comply with scheduled assessments and with management of toxicities.

Exclusion Criteria:

1. Other tumor type than adenocarcinoma (e.g. leiomyosarcoma, lymphoma) or a second cancer except in patients with squamous or basal cell carcinoma of the skin or carcinoma in situ of the cervix that has been effectively treated. Patients curatively treated for any other malignancy and disease-free for at least 5 years will be discussed with the sponsor before inclusion
2. Concurrent chronic systemic immune therapy, chemotherapy, or hormone therapy not indicated in the study protocol
3. Previous therapy with, paclitaxel or ramucirumab or pretreatment with a PD-1, PD-L1 Inhibitor
4. Current treatment with any anti-cancer therapy ≤ 2 weeks prior to study treatment start unless rapidly progressing disease is measured
5. Previous exposure to a VEGF (vascular endothelial growth factor) or VEGFR inhibitor or any antiangiogenic agent, or prior enrolment in this study
6. Major surgical procedure, open biopsy or significant traumatic injury within 4 weeks prior to start of study treatment; anticipation of need for major surgical procedure (e.g. impending bowel obstruction) during the course of the study
7. Grade 3-4 GI bleeding within 3 months prior to enrollment
8. History of deep vein thrombosis (DVT), pulmonary embolism (PE), or any other significant thromboembolism (venous port or catheter thrombosis or superficial venous thrombosis are not considered "significant") during the 3 months prior to first dose of protocol therapy
9. Cirrhosis at a level of Child-Pugh B (or worse) or cirrhosis (any degree) and a history of hepatic encephalopathy or clinically meaningful ascites resulting from cirrhosis. Clinically meaningful ascites is defined as ascites from cirrhosis requiring diuretics or paracentesis
10. Known brain or leptomeningeal metastases
11. Known prior severe hypersensitivity to investigational product or any component in its formulations, including known severe hypersensitivity reactions to monoclonal antibodies (NCI CTCAE v5.0 Grade ≥ 3)
12. Other serious illness or medical conditions prior to study drug administration

    1. Clinically significant (i.e., active) cardiovascular disease:

       cerebral vascular accident/stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (≥ New York Heart Association Classification Class II), or serious cardiac arrhythmia requiring medication
    2. Uncontrolled or poorly controlled hypertension despite optimal medical therapy
    3. Current history of chronic diarrhea
    4. Active disseminated intravascular coagulation
    5. History of gastrointestinal perforation, fistulae or any clinically relevant arterial thromboembolic event within 6 months
    6. Active infection that, in the opinion of the investigator, may increase the risk associated with study participation, study drug administration, or would impair the ability of the subject to receive study drug
    7. Hepatitis B virus (HBV) or hepatitis C virus (HCV) infection at screening (positive HBV surface antigen or HCV RNA if anti-HCV antibody screening test positive)
    8. Active autoimmune disease that might deteriorate when receiving an immuno-stimulatory agent. Patients with diabetes type I, vitiligo, psoriasis, or hypo- or hyperthyroid diseases not requiring immunosuppressive treatment are eligible.
    9. Serious or non-healing wound, ulcer, or bone fracture within 28 days prior to first dose of protocol therapy
    10. Prior organ transplantation including allogenic stem-cell transplantation
    11. Other severe acute or chronic medical conditions including immune colitis, inflammatory bowel disease, immune pneumonitis, pulmonary fibrosis or psychiatric conditions including recent (within the past year) or active suicidal ideation or behavior; or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study
13. Current use of immunosuppressive medication,

    EXCEPT for the following:
    1. intranasal, inhaled, topical steroids, or local steroid injection (e.g., intra-articular injection);
    2. steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication
    3. short term steroids to prevent chemotherapy induced Nausea
14. The patient is receiving chronic antiplatelet therapy, including aspirin, nonsteroidal anti-inflammatory drugs (NSAIDs, including ibuprofen, naproxen, and others), dipyridamole or clopidogrel, or similar agents. Once-daily aspirin use (maximum dose 325 mg/day) is permitted
15. Vaccination within 4 weeks of the first dose of avelumab and while on trial is prohibited except for administration of inactivated vaccines
16. Subjects with interstitial lung disease that is symptomatic or may interfere with the detection or management of suspected drug-related pulmonary toxicity
17. Concurrent treatment with other experimental drugs or participation in another clinical trial with any investigational drug within 30 days but at least 5 half-lives of the IMP prior to treatment start
18. Known drug abuse/ alcohol abuse
19. Persisting toxicity related to prior therapy (NCI CTCAE v. 5.0 Grade > 1); however, alopecia, sensory neuropathy Grade ≤ 2, or other Grade ≤ 2 not constituting a safety risk based on investigator's judgment are acceptable
20. Subject pregnant or breast feeding, or planning to become pregnant within 3 months after the end of Treatment
21. Subject (male or female) is not willing to use highly effective methods of contraception (per institutional standard) during treatment and for 30 days (male or female) with avelumab and 3 months with ramucirumab after the end of Treatment
22. Patients known to have a HER2 positive cancer who have not been treated already with a HER2 targeting Agent
23. Patients with a psychiatric illness or patients imprisoned or working in the Institution of the treating physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Overall Survival Rate at 6 months | 6 months
  patients alive at 6 months

SECONDARY OUTCOMES:
Overall Survival | 40 months
  patients alive using Kaplan Meyer
Overall Survival Rate at 12 months | 12 months
  patients alive at 12 months
Progression Free Survival | 40 months
  Patients showing progressive disease
Progression Free Survival Rate at 6 months according to RECIST v1.1 | 6 months
  Patients showing progressive disease at 6 months
Progression Free Survival Rate at 12 months according to RECIST v1.1 | 12 months
  Patients showing progressive disease at 12 months
Number of participants with treatment related adverse events (AE) as assessed by common toxicity criteria CTC AE v5.0 | 40 months
  Patients reported with adverse events
Number of participants to whom the treatment could me administered as planned (feasibility). | 40 months
  number of patients who received treatment
Best response according to RECIST v1.1 | 40 months
  Proportion of patients who show response
Confirmed response rate according to RECIST v1.1 | 40 months
  Proportion of patients who show confirmed response
Duration of response | 40 months
  time how long response lasts
Amount of Tumor infiltrating lymphocytes and TCRβ & IgH; clonal evolution | 40 months
  liquid biopsy and next generation sequencing
Subgroup analyses: number of participants with Programmed Death receptor Ligand 1 (PD-L1) positive tumors. | 40 months
  number of patients with PD-L1 positive tumors in pathology assessment
Progression Free Survival (PFS) according to modified RECIST | 40 months
  Proportion of patients who show progressive disease
Overall Response Rate (ORR) according to modified RECIST | 40 months
  Proportion of patients responding

CONTACTS AND LOCATIONS:
Overall Officials: Peter Thuss-Patience, MD, Principal Investigator — Charité-University Medicine (Berlin, Germany)
Locations (1):
- Charité Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Doi T, Iwasa S, Muro K, Satoh T, Hironaka S, Esaki T, Nishina T, Hara H, Machida N, Komatsu Y, Shimada Y, Otsu S, Shimizu S, Watanabe M. Phase 1 trial of avelumab (anti-PD-L1) in Japanese patients with advanced solid tumors, including dose expansion in patients with gastric or gastroesophageal junction cancer: the JAVELIN Solid Tumor JPN trial. Gastric Cancer. 2019 Jul;22(4):817-827. doi: 10.1007/s10120-018-0903-1. Epub 2018 Dec 4. PMID 30515672
- [Derived] Thuss-Patience P, Hogner A, Goekkurt E, Stahl M, Kretzschmar A, Gotze T, Stocker G, Reichardt P, Kullmann F, Pink D, Bartels P, Jarosch A, Hinke A, Schultheiss C, Paschold L, Stein A, Binder M. Ramucirumab, Avelumab, and Paclitaxel as Second-Line Treatment in Esophagogastric Adenocarcinoma: The Phase 2 RAP (AIO-STO-0218) Nonrandomized Controlled Trial. JAMA Netw Open. 2024 Jan 2;7(1):e2352830. doi: 10.1001/jamanetworkopen.2023.52830. PMID 38261316